CLINICAL TRIAL: NCT05925803
Title: A Multicenter, Randomized, Parallel-group, Double-blind,Two-arm Phase III Study to Evaluate the Safety and Efficacy of Anifrolumab Compared With Placebo in Male and Female Participants 18 to 70 Years of Age Inclusive With Systemic Sclerosis
Brief Title: Determine Effectiveness of Anifrolumab In SYstemic Sclerosis (DAISY)
Acronym: DAISY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3460C00002; 2023-505976-31 (Other: EuCTR)
Record Dates: First submitted 2023-06-02; First posted 2023-06-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Systemic Sclerosis; Scleroderma
Keywords: Systemic Sclerosis (SSc); Scleroderma; Anifrolumab; Limited; Diffuse; Cutaneous; Interstitial lung disease (ILD); Autoimmune diseases; Immune system diseases; Immunosuppressants; Systemic Sclerosis interstitial lung disease (SSc- ILD)
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Lung Diseases, Interstitial; Autoimmune Diseases; Immune System Diseases | interventions — anifrolumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to either anifrolumab or matching placebo for 52 weeks (double blind treatment period). At Week 52, all patients will be treated with Anifrolumab for 52 weeks (open label treatment period).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind period- masking -everyone will be masked to the treatment allocation during the first 52 weeks Open label period - no masking- beginning at week 52, all participants will receive Anifrolumab for 52 weeks. During the open label period, there is no masking of study treatment, however, the treatment that participants received in the double blind period (first 52 weeks) will remain masked until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anifrolumab (subcutaneous weekly injection) (Experimental): Anifrolumab subcutaneous injection once weekly
  Interventions: Combination Product: Anifrolumab (blinded); Combination Product: Anifrolumab (unblinded, open label)
- matched placebo control (subcutaneous weekly injection) (Placebo Comparator): matched placebo control subcutaneous injection once weekly
  Interventions: Drug: Placebo (blinded)

INTERVENTIONS:
Combination Product: Anifrolumab (blinded) — Anifrolumab treatment delivered subcutaneously, once weekly for 52 weeks
  Other Names: Treatment arm (blinded)
  Arms: Anifrolumab (subcutaneous weekly injection)
Drug: Placebo (blinded) — matched placebo delivered subcutaneously, once weekly for 52 weeks
  Other Names: Placebo arm (blinded)
  Arms: matched placebo control (subcutaneous weekly injection)
Combination Product: Anifrolumab (unblinded, open label) — At Week 52, all patients will receive Anifrolumab subcutaneously once weekly for 52 weeks
  Other Names: Treatment arm (not blinded)
  Arms: Anifrolumab (subcutaneous weekly injection)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of treatment with subcutaneous anifrolumab versus placebo in adult participants with systemic sclerosis. The target population for this study includes patients who meet the 2013 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) classification for systemic sclerosis, either limited or diffuse cutaneous subsets, with a disease duration of less than 6 years from first non-Raynaud's phenomenon symptom.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, Phase III study to evaluate the efficacy and safety of anifrolumab in the treatment of adult participants with Systemic Sclerosis (SSc) who may be taking one or a combination of protocol-specified standard therapies. The use of one of the following standard immunosuppressant therapies is permitted at a stable dose, but not mandated: hydroxychloroquine, mycophenolate mofetil (MMF), mycophenolic acid or mycophenolate sodium (MPA/MPS), methotrexate, azathioprine, tacrolimus, and oral glucocorticoids. MMF or MPA/MPS, azathioprine, and methotrexate may be used in combination with hydroxychloroquine and/or low-dose oral glucocorticoids [≤ 10 mg/day].

Approximately 306 eligible participants will be randomized in a 1:1 ratio to receive either anifrolumab (or matching placebo) given subcutaneously once weekly for 52 weeks. The study will be stratified by the following factors:

* Interstitial lung disease (ILD) (yes, no) at Week 0 (Day1);
* MMF or MPA/MPS use (yes ,no) at Week 0 (Day 1); and
* Disease duration, defined as the time from the first non-Raynaud's symptom attributable to SSc (<18 months, ≥ 18 months) at Week 0 (Day 1)

Study treatment will be administered subcutaneously via an accessorized prefilled syringe by study staff or by the participant or carer, either in the clinic or at home, with most doses being administered at home. The study consists of 4 periods: a 6-week screening period, a 52-week, double-blind, placebo-controlled period, a 52-week open-label active treatment period, and a 12-week safety follow-up period. There are a total of 16 study visits with most visits in the treatment period occurring every 8 to 12 weeks. The periods are described below:

* Screening Period: This may involve one or more visits to the study site.
* Double Blind Treatment Period: Treatment Period when participants will receive once weekly injections of anifrolumab or matching placebo. Participation will involve in-clinic study visits at Weeks 0 (Day 1), 1, 4, 8*, 16, 24, 36, 48 and 52. *The visit at Week 8 may be either by telephone or in person.
* Open Label Treatment Period: At Week 52, all participants will be given anifrolumab (subcutaneous) once weekly for 52 weeks (last dose at Week 103). Participation will involve in-clinic study visits at Weeks 52, 53*, 56, 64, 76. 88 and 104. *The visit at Week 53 may be either by telephone or in person.
* Safety Follow-up Period: All participants will return to the clinic for a 12-week post treatment visit. This will occur post Double Blind Treatment Period (Week 52 or Double Blind Period early discontinuation) or post Open Label Treatment Period (Week 104 or Open Label Period early discontinuation).

ELIGIBILITY:
Key Inclusion Criteria:

1. Adult patients from 18 to 70 years of age inclusive
2. Systemic sclerosis according to 2013 ACR/EULAR classification criteria
3. Limited or diffuse cutaneous subsets
4. Systemic sclerosis disease duration within 6 years from first non-Raynaud's phenomenon manifestation at the time of signing the ICF
5. Either HAQ-DI score ≥ 0.25 points or PtGA score ≥ 3 points
6. mRSS > 10 with early disease or rapid progression as defined by the protocol
7. mRSS ≥ 15 with disease duration ≥ 18 months and active disease as defined by the protocol
8. Stable background therapies can be used including hydroxychloroquine, methotrexate, azathioprine, mycophenolate mofetil, mycophenolate sodium, mycophenolic acid, oral glucocorticoids or tacrolimus
9. Women of childbearing potential with a negative urine pregnancy test
10. Uninvolved skin at injection sites

Key Exclusion Criteria:

1. Anticentromere antibody seropositivity on central laboratory
2. Severe cardiopulmonary disease as defined by the protocol
3. History of systemic sclerosis renal crisis within past 12 months (estimated glomerular filtration rate(eGFR) < 45 mL/min/1.73m2)
4. Overlap syndromes, systemic lupus erythematosus with anti-double-stranded deoxyribonucleic acid antibody seropositivity or anti-citrullinated protein antibodies-positive rheumatoid arthritis, or SSc mimics (eg, scleromyxedema, eosinophilic fasciitis)
5. History of, or current, any other inflammatory diseases, eg, inflammatory bowel disease, skin disease, that, in the opinion of the investigator, could interfere with efficacy and safety assessments or require immunomodulatory therapy
6. Evidence of moderately severe concurrent nervous system, renal, endocrine, hepatic (eg, underlying chronic liver disease [Child Pugh A, B, C hepatic impairment]), or gastrointestinal disease (eg, clinical signs of malabsorption or needing parenteral nutrition) not related to SSc, as determined by the investigator
7. Hematopoietic stem cell transplantation or solid organ/limb transplantation
8. Any severe case of Herpes Zoster infection as defined by the protocol
9. Known malignancy or a history of malignancy within 5 years, with exception of excised/cured local basal or squamous cell carcinoma of the skin or carcinoma in situ of the uterine cervix
10. Major surgery within 8 weeks prior to and/or during study enrollment
11. Known active current or history of recurrent infections
12. Any condition that, in the opinion of the investigator or AstraZeneca, would interfere with the efficacy or safety evaluation of the study intervention or put participant at safety risk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-10-09 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants responding to treatment based on the Revised Composite Response Index in Systemic Sclerosis (CRISS-25) | at Week 52
  Number of participants meeting all the criteria:
  * Improvement in at least 2 components (≥5% increase for percent predicted Forced Vital Capacity (FVC) and/or≥25% decrease for Modified Rodnan Skin Score (mRSS), Health Assessment Questionnaire Disability Index (HAQ-DI), Patient Global Assessment (PtGA), Clinician Global Assessment (CGA)
  * Worsening in no more than one component (≥5% decrease percent predicted FVC and/or≥25% increase for mRSS, HAQ-DI, PtGA, CGA)
  * No significant SSc-related event as defined by:
  New scleroderma renal crisis New decline in percent predicted FVC≥15% in established interstitial lung disease or new percent predicted FVC below 80% predicted New onset of left ventricular failure requiring treatment New onset of pulmonary arterial hypertension requiring treatment Gastrointestinal dysmotility requiring enteral or parenteral nutrition Digital ischemia with gangrene, amputation, or hospitalization requiring treatment
  -Otherwise, a participant is a non-responder

SECONDARY OUTCOMES:
Change from baseline in mRSS | at Week 52
  Change from baseline in mRSS score. The mRSS scoring ranges from 0 (normal) to 51 (severe).
Number of patients with improvement in individual revised Composite Response Index in Systemic Sclerosis (CRISS-25) | at Week 52
  Number of participants who have improvements in the following improvement components, evaluated separately:
  * ≥ 5% increase in percent predicted Forced Vital Capacity (FVC)
  * ≥ 25% decrease in mRSS
  * ≥ 25% decrease in HAQ-DI
  * ≥25% decrease in PtGA
  * ≥25% decrease in CGA
Change from baseline in chest computed tomography imaging | at Week 52
  Change from baseline in quantitative interstitial lung disease score
Change from baseline in Scleroderma Skin Patient Reported Outcome | at Week 52
  Change from baseline in the Scleroderma Skin Patient Reported Outcome scores
Change from baseline in FVC | at Week 52
  1. Change from baseline in FVC (ml) in patients with interstitial lung disease
  2. Change from baseline in FVC (ml) in all patients
Change from baseline in percent predicted FVC | at Week 52
  1. Change from baseline in percent predicted FVC in patients with interstitial lung disease
  2. Change from baseline in percent predicted FVC in all patient
Anifrolumab pharmacokinetic parameters in serum | Weeks 4, 16, 24, 36, 52, 56, 76, and 104 to follow-up (max 116 weeks)
  Anifrolumab serum concentrations will be summarised using descriptive statistics at each visit. Due to sparse pharmacokinetic sampling, the pharmacokinetic assessment will be primarily based on observed serum trough concentrations (Ctrough)
Anifrolumab pharmacodynamics via changes in type I IFN 21-gene signature generated from blood | Double-blind treatment period: pre-dose (Day 1) Weeks 4, 16, 24, 52; open-label period: weeks 56, 76 and 104
  Type I Interferon inducible gene signature will be assessed by a 21-gene assay in whole blood. The suppression of the type I IFN 21-gene signature will be showed as a percent of baseline through study completion, during both the double-blind treatment and open label periods.
Prevalence of anti-drug antibodies to Anifrolumab | Weeks 4, 16, 24, 36, 52, 56, 76, and 104 to follow-up (max 116 weeks)
  Anti-drug antibodies and titer determination in anti-drug antibody positive participants. The presence of neutralizing anti-drug antibodies will also be tested in all anti-drug positive samples.
Incidence of adverse events | From screening to follow-up (max 126 weeks)
  Adverse events (non-serious, serious, and adverse event of special interest (AESI)) are assessed as variables of safety and tolerability of anifrolumab.
  The AESIs are non-opportunistic serious infections, opportunistic infections, malignancy, herpes zoster, Tuberculosis (TB) (including latent TB), injection site reactions, and major adverse cardiac events.
Incidence of abnormal vital signs | From screening to follow-up (max 126 weeks)
  Change from baseline of pulse rate, blood pressure, respiration rate, and body temperature will be assessed by visit and treatment group including participants with treatment-emergent changes.
Incidence of abnormal laboratory parameters | From screening to follow-up (max 126 weeks)
  Changes from baseline in haematology, clinical chemistry and lipid variables will be assessed by visit and treatment including participants with treatment-emergent changes.
Incidence of abnormal ECG findings | From screening to end of treatment visit (max 110 weeks)
  Observed values of heart rate, QRS duration, PR interval, RR interval and QT interval will be summarised by visit and treatment group including participants with clinically significant abnormal results.
Incidence of abnormal physical exam findings | From screening to follow-up (max 126 weeks)
  Changes from baseline in weight (kilograms) will be assessed by visit and treatment and medically significant changes from the screening physical examination will be recorded as adverse events.
Number of subjects with suicidal ideation and behavior and suicide attempts via Columbia-Suicide Severity Rating Scale (C-SSRS) | From screening to follow-up (max 126 weeks)
  The C-SSRS is used to assess suicidal ideation, behavior, and suicide on a graded scale from 1 to 5. 1 indicates as low suicidal and 5 as high suicidal behavior.
Total score of Personal Health Questionnaire Depression Scale-8 (PHQD-8) | From screening to follow-up (max 126 weeks)
  PHQ-8 is an 8-item self-report scale, all items are rated on a score of 0-3, for a total range of 0-24. PHQD-8 assesses symptoms of depression over the previous 2 weeks. Higher scores indicate more depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (129):
- United States (26):
  - Research Site, Scottsdale, Arizona
  - Research Site, Chula Vista, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boca Raton, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Margate, Florida
  - Research Site, South Miami, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Kansas City, Kansas
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Babylon, New York
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Allen, Texas
  - Research Site, Houston, Texas
- Austria (3):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Vienna
- Belgium (2):
  - Research Site, Ghent
  - Research Site, Leuven
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec
- China (6):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Lanzhou
  - Research Site, Shanghai
  - Research Site, Tianjin
- France (6):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (5):
  - Research Site, Freiburg im Breisgau
  - Research Site, Mainz
  - Research Site, Minden
  - Research Site, Münster
  - Research Site, Tübingen
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Pécs
  - Research Site, Szeged
- India (10):
  - Research Site, Ahmedabad
  - Research Site, Delhi
  - Research Site, Gurugram
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, Mysuru
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Secunderabad
- Israel (5):
  - Research Site, Afula
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Ramat Gan
- Italy (6):
  - Research Site, Ancona
  - Research Site, Brescia
  - Research Site, Cona
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Roma
- Japan (14):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Iruma-Gun
  - Research Site, Kanazawa
  - Research Site, Maebashi
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
  - Research Site, Takatsuki-shi
  - Research Site, Toyoake-shi
  - Research Site, Yokohama
- Malaysia (3):
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
  - Research Site, Seremban
- Mexico (4):
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, San Luis Potosí City
- Research Site, Groningen, Netherlands
- Poland (5):
  - Research Site, Bydgoszcz
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Sosnowiec
  - Research Site, Warsaw
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Iași
- South Africa (2):
  - Research Site, Parktown
  - Research Site, Pretoria
- South Korea (2):
  - Research Site, Busan
  - Research Site, Seoul
- Spain (5):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Valencia
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Kazımkarabekir
  - Research Site, Kocaeli
  - Research Site, Merkez
- United Kingdom (4):
  - Research Site, Cannock
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Sheffield
- Vietnam (4):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AstraZeneca disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AstraZeneca group of companies sponsored clinical trials are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. The timelines vary per request and can take up to a year upon full submission of the request for analysis, decision, anonymisation and sharing of the requested data or documents. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved, AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home